CLINICAL TRIAL: NCT04746287
Title: First-in-Human, Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effects of CKD-510 in Single Ascending Dose and Multiple Ascending Dose in Healthy Subjects
Brief Title: Evaluation of the Safety and Tolerability of CKD-510 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A96_01CMT1914
Record Dates: First submitted 2021-01-15; First posted 2021-02-09 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Drug: CKD-510 Drug: Placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental): Single dose administration
  Interventions: Drug: CKD-510 single dose
- Part B (Experimental): Multiple dose administration (food Effect)
  Interventions: Drug: CKD-510 food effect
- Part C (Experimental): Multiple dose administration
  Interventions: Drug: CKD-510 multiple dose
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CKD-510 single dose — Investigational drug
  Arms: Part A
Drug: CKD-510 food effect — Investigational drug
  Arms: Part B
Drug: CKD-510 multiple dose — Investigational drug
  Arms: Part C
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a first-in-human study of CKD-510 in single-ascending dose and multiple-ascending dose in healthy subjects. This trial is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics of food effects of CKD-510.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Non-smoker subject or light smoker
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive at screening
* Laboratory parameters within the normal range of the laboratory.
* Male volunteers must be either vasectomized or agree to use a condom during the course of the study and until 3 months (90 days) after the participant's last visit
* Signing a written informed consent prior to selection

Exclusion Criteria:

* Any history or presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic or infectious disease
* Blood donation within 2 months before administration
* General anesthesia within 3 months before administration
* Presence or history of drug hypersensitivity, or allergic disease
* Any drug intake (except paracetamol or contraception) during the 28 days prior to the first administration
* History or presence of alcohol or drug abuse
* Subject who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development
* Use of an investigational drug within 3 months (or 90 days) prior to Day1

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
[Part A, Part C] Number of subjects with adverse events (AEs) | Treatment duration up to 4 days
  The relationship of each adverse event to the investigational product was assessed by the investigator.
[Part A, Part C] Safety as assessed by vital signs | Treatment duration up to 4 days
  Symptoms of vital signs will be assessed.
[Part A, Part C] Safety as assessed by abbreviated physical examination parameters | Treatment duration up to 4 days
  Physical exmaination will include evaluation of main body systems/regions
[Part A, Part C] Safety as assessed by electrocardiogram (ECG) parameters | Treatment duration up to 4 days
  12-lead ECGs will be obtained during the study using an ECG machine
[Part A, Part C] Safety as assessed by biological analysis | Treatment duration up to 4 days
  Biological test will be obtained with assessments including hematology, biochemistry, urinalysis.
[Part B] Composite of pharmacokinetics (PK) assessments of CKD-510 | 3 days post dose
  PK parameters include plasma concentrations of CKD-510, maximum observed plasma concentration (Cmax), time to Cmax (tmax), area under the plasma concentration-time curve (AUC) to last measurable concentration [AUC(0-t)], AUC through 24 hours [AUC(0-24)] and AUC per dosing interval [AUC(0-tau)], apparent terminal phase half-life following the last dose (t1/2) in fast or fed conditions.
[Part B] Composite of pharmacodynamics (PD) assessments of CKD-510 | 3 days post dose
  Change from baseline in acetylation of alpha-tubulin and histone as pharmacodynamics assessments after an administration of CKD-510 in fast or fed conditions

SECONDARY OUTCOMES:
[Part A, Part C] Maximum plasma concentration of CKD-510 | 4 days post dose (SAD) or 17 days post dose (MAD)
  Peak plasma concentration (Cmax)
[Part A, Part C] Time of maximum plasma concentration of CKD-510 | 4 days post dose (SAD) or 17 days post dose (MAD)
  Time to reach Cmax (Tmax)
[Part A, Part C] Changes from baseline in plasma concentrations CKD-510 in time after dosing | 4 days post dose (SAD) or 17 days post dose (MAD)
  Area under the concentration-time curve from time 0 extrapolated to the last quantifiable concentration at time t (AUC0-t)
[Part A, Part C] Time of plasma elimination half-life of CKD-510 | 4 days post dose (SAD) or 17 days post dose (MAD)
  Apparent terminal elimination half-life (t½)
[Part A, Part C] Volume of distribution of CKD-510 | 4 days post dose (SAD) or 17 days post dose (MAD)
  Apparent volume of distribution during the terminal elimination phase (Vd/F)
[Part A, Part C] Total plasma clearance of CKD-510 | 4 days post dose (SAD) or 17 days post dose (MAD)
  Apparent total plasma clearance (CL/F)
[Part A, Part C] Pharmacodynamics assessments of CKD-510 | up to 2 days post dose (SAD) or 17 days post dose (MAD)
  Change from baseline in acetylation of alpha-tubulin and histone
[Part B] Number of subjects with adverse events (AEs) | 3 days post dose
  The relationship of each adverse event to the investigational product was assessed by the investigator
[Part B] Safety as assessed by vital signs | 3 days post dose
  Symptoms of vital signs will be assessed.
[Part B] Safety as assessed by abbreviated physical examination parameters | 3 days post dose
  Physical exmaination will include evaluation of main body systems/regions
[Part B] Safety as assessed by electrocardiogram (ECG) parameters | 3 days post dose
  12-lead ECGs will be obtained during the study using an ECG machine
[Part B] Safety as assessed by biological analysis | 3 days post dose
  Biological test will be obtained with assessments including hematology, biochemistry, urinalysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical site, Grenoble, France